CLINICAL TRIAL: NCT02970188
Title: The Effect of Time-restricted Feeding on Physiological Function in Middle-aged and Older Adults
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Principal Investigator, Douglas Seals, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15-0108
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Aging
Keywords: time restricted feeding; endothelial function; arterial stiffness; intermittent fasting
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Feeding (No Intervention): Subjects will be instructed to eat within their normal feeding window.
- Time Restricted Feeding (Experimental): Subjects will be instructed to eat with an 8 hour feeding window, starting between 10:30-11:30 AM and stopping between 5:30-6:30 PM.
  Interventions: Behavioral: Time Restricted Feeding

INTERVENTIONS:
Behavioral: Time Restricted Feeding — consuming all daily calories within an 8 hour feeding window
  Other Names: TRF
  Arms: Time Restricted Feeding

SUMMARY:
The purpose of this study is to assess the safety and efficacy of time-restricted feeding (eating within an 8-hour window) for improving physiological function (vascular, motor, cognitive and metabolic function) in healthy middle-aged and older adults.

DETAILED DESCRIPTION:
Overall, the proposed research project has the long-term potential to influence clinical practice by establishing novel therapies for treating multiple domains of age-associated physiological dysfunction and thereby reducing the risk of clinical disease and disability.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Baseline brachial flow-mediated dilation (FMD) < 6%Δ (rationale: non-invasive screening to ensure exclusion of subjects with exceptionally high baseline endothelial function.
* Ability to perform motor and cognitive tests (e.g., can rise from a chair, walk for 2 min, climb 10 stairs)
* Women will be confirmed as postmenopausal (either natural or surgical) based on cessation of menses for >1 year.

Exclusion Criteria:

* Ages <55 years or ≥80 years
* Occupation that requires night-shift work or abnormal hours that would disrupt eating schedule
* Dietary habit of regularly skipping meals, already eating within a ~10 hour window, or any other form of restrictive eating.
* Unable to adhere to an 8 hour eating window for the length of the study period
* Participation in regular vigorous aerobic/endurance exercise (>3 vigorous bouts/week)
* Not weight stable in the prior 3 months (>2 kg weight change).
* Body mass index (BMI) >40 kg/m^2 (rationale: vascular function measurements can be inaccurate in severely obese subjects)
* Current smoking
* Diagnosis of a chronic clinical disease (e.g., coronary artery/peripheral artery/cerebrovascular diseases, diabetes, chronic kidney disease requiring dialysis, neurological disorders or diseases that may affect motor/cognitive functions [multiple sclerosis, Parkinson's disease, polio, Alzheimer's disease, dementia or other brain diseases of aging]), except hypertension and hyperlipidemia.
* Having unstable angina, acute myocardial infarction, coronary angioplasty, or aorto- coronary bypass surgery as defined by the occurrence of an event, symptom, surgery, or change in medication and/or dosage within 3 months prior to enrollment.
* Having thyroid disease that is not controlled by medications or <3 month's use of a particular medication and/or dosage (rationale: uncontrolled thyroid diseases are associated with alterations in vascular function).
* Having past or present alcohol dependence or abuse, as defined by the American Psychiatry Association, Diagnostic and Statistical Manual of Mental Disorders

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-01 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Endothelium Dependent Dilation | 6 weeks
  Brachial Artery Flow-Mediated Dilation (FMD)

SECONDARY OUTCOMES:
Arterial Stiffness | 6 weeks
  Aortic Pulse Wave Velocity (PWV)
Cognitive Function | 6 weeks
  NIH Toolbox Cognitive Function Battery
Motor Function | 6 weeks
  NIH Toolbox Motor Function Battery
Metabolic Function | 6 weeks
  Oral glucose tolerance test (OGTT)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R Martens, Ph.D., Principal Investigator — University of Colorado, Boulder
Locations (1):
- Integrative Physiology of Aging Laboratory, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717